CLINICAL TRIAL: NCT03796663
Title: Evaluation of the Effectiveness of a Combined Mindful Parenting and Parent Training Program on Children With Disruptive Behavioral Problems and Their Families
Brief Title: Mindful Parenting and Parent Training Program Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2019-2401
Record Dates: First submitted 2018-12-19; First posted 2019-01-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2021-06

CONDITIONS: Disruptive Behavior; Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder; Conduct Disorder; Disruptive Behavior Disorder
Keywords: Disruptive Behavioral Problems; ADHD; Oppositional Defiant Disorder; Conduct Disorder; Mindfulness; Mindful Parenting; Behavioral Parent Training
MeSH Terms: conditions — Problem Behavior; Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Intervention Model Description: All participants will receive the Mindful Parenting program at the start of their involvement in the study. Following the completion of the Mindful Parenting group sessions, half of the participants will be randomly selected to receive individually-implemented MATCH BPT sessions. The other half of families will have the opportunity to also receive the MATCH BPT program following the completion of data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Parenting Only (Active Comparator): Participants in this arm will receive only the Mindful Parenting Program at the start of the study. Bögels and Restifo's (2014) Mindful Parenting Program is an adaptation for parents of MBCT, and MBSR; the program will consist of 7-weekly 2.5-hour parent group sessions. In the program, parents learn to apply the skills of mindfulness to themselves and to their experience of parenting their children.
  Following the completion of the Mindful Parenting Sessions, participants in this arm will be asked continue to participate in data collection for the post-intervention assessment time point (i.e. 8 weeks after the completion of the Mindful Parenting group sessions) and for the 2-month follow up assessment time point (i.e. 16 weeks after the completion of the Mindful Parenting group sessions). After they have completed both assessments, they will be offered the opportunity to participate in the MATCH BPT program if they so choose (no data will be collected).
  Interventions: Behavioral: Mindful Parenting Program
- Mindful Parenting and BPT Combined (Experimental): Participants in this arm will receive the Mindful Parenting Program at the start of the study, which will consist of 7-weekly 2.5-hour parent group sessions. In the program, parents learn to apply the skills of mindfulness to themselves and to their experience of parenting their children.
  Following the completion of the Mindful Parenting Sessions, participants in this arm will receive receive individually-implemented MATCH BPT sessions, which will consist of 8-12 weekly (depending on how long it takes for individual parents and their assigned trainer to get through the material), 1 hour sessions. The MATCH manual is comprised of 33 modules (i.e. coping, giving effective instructions, learning to relax, etc.). For the purpose of this study we will be utilizing the section on BPT, which consists of 12 modules with corresponding handouts and worksheets.
  Interventions: Behavioral: Mindful Parenting Program; Behavioral: MATCH BPT Program

INTERVENTIONS:
Behavioral: Mindful Parenting Program — The Mindful Parenting Program consists of 7, 2.5 hour weekly group sessions. In the program, parents learn to apply the skills of mindfulness to themselves and to their experience of parenting their children. Parents are introduced to formal meditation practices, including the bodyscan; choiceless awareness; mindful walking; and yoga. They are also introduced to mindfulness of everyday activities from the beginning of the sessions, with an added focus on day-to-day parenting and family activities. Additionally, short self-compassion practices occur throughout the weekly sessions, culminating in the teaching of formal loving-kindness meditation.
  Additionally, the program encourages parents to engage in "home practice", where parents can experience and practice many of the new skills they are learning. This includes both formal, longer meditation practices, as well as shorter practices, which can occur throughout the day, such as mindfulness of daily routines.
Behavioral: MATCH BPT Program — The MATCH BPT Program consists of 8-12 weekly (depending on how long it takes for individual parents and their assigned trainer to get through the material), 60 minute individually-implemented sessions.The sessions will consist of the coach obtaining and reviewing weekly assignments completed by the parent, followed by activities and discussions that focus on a particular parenting skill (i.e. praise, active ignoring, giving effective instructions). The discussions will emphasize benefits and possible problems that the parent may encounter throughout the week while implementing the new skill. The coach will assign to the parent a practice assignment to further encourage use of the concept.
  Arms: Mindful Parenting and BPT Combined

SUMMARY:
The Mindful Parenting and Parent Training Study will be investigating the combination of Bögels and Restifo's (2014) Mindful Parenting Program and Chorpita and Weisz's (2009) Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems (MATCH) Program, specifically the BPT module. The Mindful Parenting Program is an adaptation for parents of the Mindfulness-Based Cognitive Therapy, and the Mindfulness-Based Stress Reduction program; the program will consist of 7-weekly 2.5-hour parent group sessions. Following the completion of the Mindful Parenting group sessions, half of the participants will be randomly selected to receive individually-implemented MATCH BPT sessions, which will consist of 8-12 weekly (depending on how long it takes for individual parents and their assigned trainer to get through the material), 1.5-hour sessions. The other half of families will have the opportunity to also receive the MATCH BPT program following the completion of data collection.

Both evaluation and treatment services will be offered at no cost to study participants. Parents, children, and teachers will also be offered monetary incentive to thank them for their time and effort completing study related assessments throughout the course of the study to determine if the combination of the Mindful Parenting Program with BPT improves functioning in children with disruptive behavioral problems, as well as the parent-child relationship and the parent's acquisition and enactment of the skills they learn in BPT.

ELIGIBILITY:
Inclusion Criteria:

1. the child participant must be between the ages of 6 and 11 years old at baseline/time of pretreatment data collection;
2. he/she must have an elevated score (i.e. a t-score of 60 or greater) on one or more of the Externalizing Problems clinical scales (i.e. Hyperactivity, Aggression, and Conduct Problems) or on the Attention Problems clinical scale of the Behavior Assessment System for Children 3rd Edition - Parent Report (BASC-3; Reynolds & Kamphaus,

2015), as assessed during the intake assessment for the study; 3) both the parent and child participants must be fluent English speakers, and; 4) the parent participant(s) must be available to attend weekly treatment sessions and assessments for up to 26 weeks at New York University - Kimball Hall.

Exclusion Criteria:

1. There is evidence of significant developmental delay or psychosis that impacts the child's ability to fully engage in the intervention;
2. The youth or parent presents with emergency psychiatric needs that require services beyond that which can be managed within this intervention format (e.g. hospitalization, specialized placement outside the home);
3. if the parent and/or child are not fluent English speakers;
4. if the family is currently enrolled in any type of behavioral parent or parent management training program; and
5. if the child has an estimated Full Scale IQ below 80, based on completing two subtests of the Wechsler Abbreviated Scale of Intelligence, Second Edition during the intake assessment for the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Behavioral Assessment System for Children - 3 (BASC-3) | Seven months from start of intervention.
  A well-standardized, multidimensional approach to evaluating the behavior of children. For this measure we will be looking at several subscales, including Hyperactivity, Agression, Conduct Problems, Externalizing Problems, Attention Problems, Anger Control, and Emotional Self-Control. For each subscale, a T-score is obtained using norms; T-scores range from 20 to 120, with higher T-Scores indicating a worse outcome/greater impairment.
Brief Problem Checklist-Parent (BPC-P) | Seven months from start of intervention.
  A measure designed to periodically assess the clinical progress of a child over the course of psychological treatment, specifically measuring the severity of internalizing and externalizing problems found in children. The scale scores of the BPC are based on the raw sum of item responses, each of which ranges from 0 to 2. Thus, scores on the six-item Internalizing and Externalizing scales each range from 0 to 12, and scores on the Total Problems scale range from 0 to 24, with higher scores indicating increased problem levels.
Impairment Rating Scale - Parent/Teacher Version (IRS) | Seven months from start of intervention.
  A multidimensional measure that assesses functioning across domains. Specifically, the IRS qualifies and quantifies impairment present in a child's life, both in school and non-school settings. No total or subscale scores are calculated, each item of this measure is considered individually.
Columbia Impairment Scale (CIS) | Seven months from start of intervention.
  Measures 4 major areas of functioning: interpersonal relations, broad psychopathological domains, functioning in job or schoolwork, and use of leisure time. Items are scored on a 5-point Likert-type scale ranging from 0 ("no problem") to 4 ("a very big problem"). "Not applicable/do not know" is scored as a 5. Sum scores can range from 0 to 52, with higher scores indicating greater impairment.
Mindfulness In Parenting Questionnaire (MIPQ) | Seven months from start of intervention.
  Assesses two factors of mindfulness in parenting: Being in the moment with the child and mindful discipline. For all 28 items, parents rate themselves for each item using the following scale: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = almost always. Standard Scores are obtained for each subscale by summing up the items that make up that subscale and then using a conversion table.
Five-Facet Mindfulness Questionnaire (FFMQ) | Seven months from start of intervention.
  A widely used scale to assess the tendency to be mindful in daily life.The FFMQ is a 39-item self-report measure that evaluates five facets of the tendency to be mindful in daily life and consists of the five subscales of Observing (scores range from 8 to 40), Describing (scores range from 8 to 40), Acting with Awareness (scores range from 8 to 40), Nonreactivity (scores range from 7 to 35), and Nonjudging (scores range from 8 to 40). The scale uses a five-point Likert scale for all items, where 1 = never or very rarely true and 5 = very often or always true. For all subscales a higher score is indicative of a greater tendency to be mindful in that particular facet. The two subscales are Mindful Discipline and Being in the Moment with the Child; for both scales, Standard scores between 90 and 110 fall within the average range, with higher scores indicating greater levels of mindful parenting.
Parent-Child Interaction Questionnaire-Revised-Parent and Child Version (PACHIQ-R) | Seven months from start of intervention.
  Assesses how parents view their relationship with their children (and how children view their relationship with their parents). There are 25 items split into two parts, part 1 with items 1 through 14 and part 2 with items 15 through 25 in the PACHIQ-R questionnaire. The Total Score ranges from 25 to 125. A high Total Score is indicative for a positive relationship.
Parenting Scale (PS) | Seven months from start of intervention.
  Self-report measure of dysfunctional parenting in discipline situations. The measure consists of 30 items, and each item receives a 1-7 score. The Total Score is calculated by averaging the responses on all 30 items and ranges from 1 to 7. There are 4 subscales - Laxness, Overreactivity, Verbosity, and Other - the scores for which are also calculated by averaging the responses on the items that make up each subscale. The score for each subscale ranges from 1 to 7. For each score, lower numbers indicate a higher probability of using effective discipline strategies and higher numbers indicate a higher probability of using ineffective discipline strategies.
Parent Behavior Inventory (PBI) - Supportive/Engaged Subscale | Seven months from start of intervention.
  Measure of parenting behavior that contains two independent scales, Supportive/Engaged and Hostile/Coercive. We will only be looking at the Supportive/Engaged Subscale, which measures levels of supportive/engagement parenting behavior. For this subscale, parents rate themselves for each item using the following scale: 0 = not at all true, 1 = a little true, 2 = somewhat true, 3= moderately true, 4 = quite a bit true, 5 = very true. To obtain To obtain the Subscale score, the responses to each item are summed together; the score can range from 0 to 50. A higher score is indicative of parents engaging in more supportive or engaged parenting behaviors.
Family and Peer Process Code (FPP) and Five Observational Lab Tasks | Seven months from start of intervention.
  Parenting practices will be assessed using data derived from 35 min of videotaped parent-child interaction. These interactions will sample five different tasks. Trained observers blind to intervention assignment will then code the tapes of the family interaction using the FPP and will make global ratings.
IOWA Conners Rating Scale | Seven months from start of intervention.
  The first half of the measure is designed to assess inattentive-impulsive-overactive behaviors while the second half captures behaviors related to oppositional-defiant activity. All 10 items of the measure are scored using a four point Likert scale with the following anchors: not at all (0); just a little (1); pretty much (2); and very much (3). The first five items on the IOWA are designed to measure inattentive-impulsive-overactive (IO Subscale) behaviors and the second five items are designed to measure oppositional-defiant (OD Subscale) behaviors. For both scales, higher scores indicate greater impairment and the scores can range from 0 to 15.

SECONDARY OUTCOMES:
Parent Emotion Regulation Inventory-2 (PERI-2) | Seven months from start of intervention.
  Measures parent emotions and their ability to regulate their emotions during interactions with their child. This measure consists of items, on which parents rate themselves for each item using a Likert scale of 1 (I never do this) to 7 (I very often do this). We will be looking at two subscales - Reappraisal and Suppression; the scores for both subscales are calculated by taking the average of the responses on the items for each subscale, and so each of the subscales scores can range from 1 to 7. For the Reappraisal scale, a higher score indicates a more frequent use of reappraisal as an emotional regulation strategy, and for the Suppression Subscale a higher score indicates a more frequent use of suppression as an emotion regulation strategy.
Knowledge of Parenting Strategies Scale (KoPSS) | Seven months from start of intervention.
  A measure of parents' knowledge of effective parenting strategies.This measure consists of 33 items, and we will be looking at the total number of correct answers obtained by the participant. As such, the score can range from 0 to 33, with a higher score indicate a greater knowledge of parenting strategies.
Emotion Regulation Questionnaire (ERQ) | Seven months from start of intervention.
  Assesses individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression. The ERQ is a 10-item scale on which parents rate each item using a Likert scale of 1 (Strongly disagree) to 7 (strongly agree). There are two subscales, Reappraisal (ranges from 1 to 42) and Suppression (ranges from 4 to 28). For the Reappraisal scale higher scores indicate a more frequent use of reappraisal as an emotional regulation strategy, and for the Suppression Subscale higher scores mean a more frequent use of suppression as an emotion regulation strategy.
Berkeley Expressivity Questionnaire (BEQ) | Seven months from start of intervention.
  A measure of parent emotional expression in discipline specific situations; it will be modified to reflect parents' emotional expression when faced with child misbehavior. We will be looking at the Total Score (which ranges from 16 to 112), as well as several subscale scores: Negative Expressivity (ranges from 6 to 42), Positive Expressivity (ranges from 4 to 28), and Impulse Strength (ranges from 6 to 42). For all scales a higher score means a greater amount of emotional expressivity is displayed by the individual.
Positive and Negative Affect Scale (PANAS) | Seven months from start of intervention.
  A measure of parent's emotional experience in discipline specific situations. The measure consists of 20 items, on which parents rate themselves for each item using the following scale: 1 = very slightly or not at all, 2 = a little, 3 = moderately, 4 = quite a bit, and 5 = very much. To calculate the Positive Affect Subscale Score, the scores on the ten items that make up the subscale are summed together. Scores can range from 10-50, with higher scores representing higher levels of positive affect. To calculate the Negative Affect Subscale Score, the scores on the 10 items that make up that subscale are summed together. Scores can range from 10-50, with lower scores representing lower levels of negative affect.
Parenting Stress Index-Short Form (PSI-SF) | Seven months from start of intervention.
  Measures the level of stress in the parent-child relationship and is appropriate for use with children aged 1 month to 12 years. It consists of 36 statements, each rated on a 1 to 5 scale (i.e., strongly disagree, disagree, not sure, agree, and strongly agree), which produces a Total Stress score that ranges from 36 to 180, with a higher score indicating greater levels of parenting stress.
Fragile Families Aggravation in Parenting Scale | Seven months from start of intervention.
  The scale measures the amount of parenting stress brought on by changes in employment, income or other factors in the parent's life. This questionnaire consists of 4 items on a Likert Scale. Parents rate themselves for each item using the following scale on a: 1 = Strongly agree, 2 = Somewhat agree, 3 = Somewhat disagree, and 4 = Strongly disagree. A Total Score is calculated by using the sum of all items divided by the top value of the Likert scale (i.e. 4); as such the Total Score ranges from 1 to 4, with a higher score indicating greater levels of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University - Kimball Hall, New York, New York, United States

REFERENCES:
- See also: FACES Lab - Study Website — https://steinhardt.nyu.edu/appsych/faceslab/